CLINICAL TRIAL: NCT03531281
Title: A Randomized Pilot Study of Human Lysozyme Goat Milk in Recipients of Standard Myeloablative Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Human Lysozyme Goat Milk in Treating Patients With Blood Cancer Undergoing Donor Stem Cell Transplant
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Administratively withdrawn
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17399; NCI-2018-00053 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17399 (Other: City of Hope Medical Center)
Record Dates: First submitted 2018-01-26; First posted 2018-05-21 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Hematopoietic Cell Transplantation Recipient
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Cyclophosphamide; Etoposide; Fibroblast Growth Factor 7; Sirolimus; Tacrolimus; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (goat milk, transplant conditioning/prophylaxis) (Experimental): CONDITIONING: Patients receive palifermin on days -10 to -8 and days 0 to 2, undergo FTBI on days -7 to -4, and receive cyclophosphamide on days -3 to -2 or etoposide on day -3 per COH SOP in the absence of disease progression or unacceptable toxicity.
  HLZ: Patients receive human lysozyme goat milk PO TID on days -8 to 28 in the absence of disease progression or unacceptable toxicity.
  TRANSPLANT: Patients undergo stem cell infusion on day 0.
  GVHD PROPHYLAXIS: Beginning on day -2, patients receive tacrolimus and sirolimus daily per COH SOP in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Cyclophosphamide; Drug: Etoposide; Drug: Goat Milk; Other: Laboratory Biomarker Analysis; Biological: Palifermin; Drug: Sirolimus; Drug: Tacrolimus; Radiation: Total-Body Irradiation
- Arm II (transplant conditioning/prophylaxis) (Active Comparator): CONDITIONING: Patients receive palifermin on days -10 to -8 and days 0 to 2 per COH SOP, undergo FTBI on days -7 to -4, and receive cyclophosphamide on days -3 to -2 or etoposide on day -3 per COH SOP in the absence of disease progression or unacceptable toxicity.
  TRANSPLANT: Patients undergo stem cell infusion on day 0.
  GVHD PROPHYLAXIS: Beginning on day -2, patients receive tacrolimus and sirolimus daily per COH SOP in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Cyclophosphamide; Drug: Etoposide; Other: Laboratory Biomarker Analysis; Biological: Palifermin; Drug: Sirolimus; Drug: Tacrolimus; Radiation: Total-Body Irradiation

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allo-HCT
  Other Names: Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Drug: Goat Milk — Given human lysozyme goat milk PO
  Arms: Arm I (goat milk, transplant conditioning/prophylaxis)
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Palifermin — Given IV
  Other Names: Growth Factor, Recombinant Human Keratinocyte; Kepivance; Keratinocyte Growth Factor, Recombinant Human; Recombinant Human Keratinocyte Growth Factor; rhKGF; rhu Keratinocyte Growth Factor
Drug: Sirolimus — Given PO
  Other Names: AY 22989; RAPA; Rapamune; Rapamycin; SILA 9268A; WY-090217
Drug: Tacrolimus — Given IV and PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic
Radiation: Total-Body Irradiation — Undergo FTBI
  Other Names: Total Body Irradiation; Whole-Body Irradiation

SUMMARY:
This randomized pilot phase I trial studies the side effects of human lysozyme goat milk in treating patients with blood cancer undergoing a donor stem cell transplant. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells (called graft-versus-host disease). Giving human lysozyme goat milk to patients undergoing a donor stem cell transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and feasibility of human lysozyme goat milk (hLZ) treatment by assessing type, frequency, severity, attribution, time course and duration of adverse events, including diarrhea, bloodstream/intestinal infections.

II. To evaluate the safety and feasibility of hLZ treatment by assessing patient compliance, the patients' ability to drink the specified volume (250 ml 3 x/day) of hLZ during the treatment period.

SECONDARY OBJECTIVES:

I. To compare the incidence and severity of adverse events (AE) among hLZ-treated and untreated patients, including diarrhea, bloodstream infections and intestinal infections.

II. To obtain preliminary estimates of gut microbiome diversity, as assessed by the Simpson Index, in hLZ-treated/untreated patients.

III. To compare gut microbiome diversity among hLZ-treated/untreated patients. IV. To obtain a preliminary estimate of the possible association between gut microbiome diversity and bloodstream infections.

V. To obtain a preliminary estimate of the possible association between gut microbiome diversity and acute graft versus host disease (GVHD) cumulative incidence, including time to onset.

VI. To characterize and compare GVHD inflammatory biomarkers (presence, level) among hLZ-treated and untreated patients.

VII. To characterize and compare urinary uindoxyl sulfate, tryptophan and kynurenine levels between hLZ-treated and untreated patients.

IX. To estimate overall survival (OS) cumulative incidence (CI) chronic GVHD of relapse/progression, and non-relapse mortality (NRM) at 100 days (excluding chronic GVHD), 6 months, 1 year and 2 years.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I:

CONDITIONING: Patients receive palifermin on days -10 to -8 and days 0 to 2, undergo fractionated total body irradiation (FTBI) on days -7 to -4, and receive cyclophosphamide on days -3 to -2 or etoposide on day -3 per City of Hope (COH) standard operating procedure (SOP) in the absence of disease progression or unacceptable toxicity.

HLZ: Patients receive human lysozyme goat milk orally (PO) three times daily (TID) on days -8 to 28 in the absence of disease progression or unacceptable toxicity.

TRANSPLANT: Patients undergo stem cell infusion on day 0.

GVHD PROPHYLAXIS: Beginning on day -2, patients receive tacrolimus and sirolimus daily per COH SOP in the absence of disease progression or unacceptable toxicity.

ARM II:

CONDITIONING: Patients receive palifermin on days -10 to -8 and days 0 to 2 per COH SOP, undergo FTBI on days -7 to -4, and receive cyclophosphamide on days -3 to -2 or etoposide on day -3 per COH SOP in the absence of disease progression or unacceptable toxicity.

TRANSPLANT: Patients undergo stem cell infusion on day 0.

GVHD PROPHYLAXIS: Beginning on day -2, patients receive tacrolimus and sirolimus daily per COH SOP in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Willingness to be followed for the planned duration of the trial (2 years)
* All subjects must have the ability to understand and the willingness to sign a written informed consent
* Karnofsky performance status >= 60 per COH SOP
* Patients must be undergoing allogeneic hematopoietic stem cell transplantation (alloHCT) for hematologic malignancies from matched related or matched unrelated donors with 8/8 (A, B, C, DRB 1) high resolution human leukocyte antigen (HLA) donor allele matching
* Patients must be receiving a fractionated total body radiation (FTBI) based- myeloablative conditioning regimen; (acceptable conditioning regimens include total body irradiation [TBI] + cyclophosphamide or TBI + etoposide)
* Ejection fraction measured by echocardiogram or multi gated acquisition scan (MUGA) > 45%
* Diffusing capacity for carbon monoxide (DLCO) adjusted for hemoglobin or forced vital capacity (FVC) > 50% predicted
* Total serum bilirubin < 2 times upper limit of normal
* Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) =< 2.5 x the upper normal limit
* Alkaline phosphatase =< 2.5 x the upper normal limit
* Measured creatinine clearance more than 60 mL/min; the updated Schwartz formula should be used for pediatric patients (>= 5 to 12 years old)
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through 90 days after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Failure of research participant to understand the basic elements of the protocol and/or the risks/benefits of participating in this pilot study; a legal guardian may substitute for the research participant
* Research participants receiving any other investigational agents
* Research participants with presence of other active malignancy within 2 years of study entry; participants with history of prior malignancy treated with curative intent who achieved complete remission (CR) more than 2 years before study entry are eligible; this exclusion rule does not apply to non-melanoma skin tumors and in-situ cervical cancer
* Research participants having any uncontrolled illness including ongoing or active infection; research participants with known active hepatitis B or C infection; research participants who are human immunodeficiency virus (HIV) seropositive based on testing performed within 4 weeks of enrollment; research participants with any signs or symptoms of active infection, positive blood cultures, or radiological evidence of infections
* Refusing to use contraception up to 90 days post-HCT
* Pregnant and/or breast feeding if a female recipient
* Lactose intolerance or intolerance to milk products
* In the opinion of the principal investigator (PI), the participant has a condition that will preclude them from complying with study treatment

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-30 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of drinking human lysozyme goat milk (hLZ) | Up to +28 days post-transplant or date of discharge
  Feasibility of drinking hLZ will be evaluated by assessment of patients' ability to drink the specified volume (250 ml 3 x per day) of hLZ during the safety lead-in phase.
Unacceptable toxicity | Up to 28 days post-transplant or date of discharge
  The modified Bearman Scale will be used to define unacceptable toxicity events. Unacceptable toxicity in a given patient is defined as either of the following that are considered at least possibly related to drinking hLZ milk: GI toxicity grade III or IV per Bearman scale or inability to consume hLZ milk for >7 days.
Adverse events | Up to 100 days post-transplant
  Incidence and severity of adverse events will be reported according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.03. Observed toxicities will be summarized in terms of type (organ affected or laboratory determination), severity, time of onset, duration, probable association with the study treatment and reversibility or outcome.
Volume of hLZ consumed | Up to 28 days post-transplant or date of discharge
  Tolerability is defined as the ability to consume >= 150 ml/day over the treatment period.

SECONDARY OUTCOMES:
Cumulative incidence (CI) of chronic GVHD | At 6 months
  Chronic graft versus host disease is scored according to NIH Consensus Staging. The first day of chronic GvHD onset will be used to calculate CI incidence curves, with relapse/death prior to onset considered competing events. CI of chronic GVHD will be estimated using the method described by Gooley et al (1999).
Cumulative incidence (CI) of chronic GVHD | At 1 year
  Chronic graft versus host disease is scored according to NIH Consensus Staging. The first day of chronic GvHD onset will be used to calculate CI incidence curves, with relapse/death prior to onset considered competing events. CI of chronic GVHD will be estimated using the method described by Gooley et al (1999).
Cumulative incidence (CI) of chronic GVHD | At 2 years
  Chronic graft versus host disease is scored according to NIH Consensus Staging. The first day of chronic GvHD onset will be used to calculate CI incidence curves, with relapse/death prior to onset considered competing events. CI of chronic GVHD will be estimated using the method described by Gooley et al (1999).
CI of non-relapse mortality (NRM) | At 100 days
  Non-relapse mortality (NRM) is defined as death occurring in a patient from causes other than relapse. NRM is measured from start of treatment until non-disease related death, or last follow-up, whichever comes first. The cumulative incidence of NRM will be calculated reflecting relapse as a competing risk. CI of NRM will be estimated using the method described by Gooley et al (1999).
CI of NRM | At 1 year
  Non-relapse mortality (NRM) is defined as death occurring in a patient from causes other than relapse. NRM is measured from start of treatment until non-disease related death, or last follow-up, whichever comes first. The cumulative incidence of NRM will be calculated reflecting relapse as a competing risk. CI of NRM will be estimated using the method described by Gooley et al (1999).
CI of NRM | At 2 years
  Non-relapse mortality (NRM) is defined as death occurring in a patient from causes other than relapse. NRM is measured from start of treatment until non-disease related death, or last follow-up, whichever comes first. The cumulative incidence of NRM will be calculated reflecting relapse as a competing risk. CI of NRM will be estimated using the method described by Gooley et al (1999).
CI of relapse/progression | At 100 days
  The event is relapse/progression. Time to this event is measured from start of treatment. Death without relapse/progression is considered a competing risk. Surviving patients with no history of relapse are censored at time of last follow-up. CI of relapse/progression will be estimated using the method described by Gooley et al (1999).
CI of relapse/progression | At 1 year
  The event is relapse/progression. Time to this event is measured from start of treatment. Death without relapse/progression is considered a competing risk. Surviving patients with no history of relapse are censored at time of last follow-up. CI of relapse/progression will be estimated using the method described by Gooley et al (1999).
CI of relapse/progression | At 2 years
  The event is relapse/progression. Time to this event is measured from start of treatment. Death without relapse/progression is considered a competing risk. Surviving patients with no history of relapse are censored at time of last follow-up. CI of relapse/progression will be estimated using the method described by Gooley et al (1999).
Gut microbiome diversity | Day - 8 +/- 3, Day 0, Day +7, Day +14, Day +21, Day +28
  Gut microbiome diversity will be assessed by the Simpson Index and compared between hLZ-treated/untreated patients. Association between treatment and gut microbial diversity will be assessed by Fisher's Exact test.
CI of acute graft versus host disease (aGVHD) | At 100 days
  Acute graft versus host disease will be graded according to the Consensus Grading. The first day of acute GvHD onset at a certain grade will be used to calculate cumulative incidence curves for that GvHD grade; relapse/death prior to onset will be considered competing events. CI of aGVHD will be estimated using the method described by Gooley et al (1999). Association between gut microbial diversity (inverse Simpson index: high [>4], intermediate [2-4], and low [<2]) or treatment and CI of aGVHD will be assessed by Gray's test.
Incidence of bloodstream infections | Up to 100 days
  Incidence of bloodstream infections and infectious enterocolitis will be evaluated and a preliminary estimate of the association between gut microbiome diversity and bloodstream infections will be obtained. Association between gut microbial diversity (inverse Simpson index: high [>4], intermediate [2-4], and low [<2]) or treatment and CI of bloodstream infections will be assessed by Gray's test.
Overall survival (OS) | At 100 days
  Patients are considered a failure for this endpoint if they die, regardless of cause. The time to this event is the time from start of treatment until death, or last follow-up, whichever comes first. OS will be estimated using the product-limit method of Kaplan and Meier.
Overall survival (OS) | At 1 year
  Patients are considered a failure for this endpoint if they die, regardless of cause. The time to this event is the time from start of treatment until death, or last follow-up, whichever comes first. OS will be estimated using the product-limit method of Kaplan and Meier.
Overall survival (OS) | At 2 years
  Patients are considered a failure for this endpoint if they die, regardless of cause. The time to this event is the time from start of treatment until death, or last follow-up, whichever comes first. OS will be estimated using the product-limit method of Kaplan and Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Karamjeet Sandhu, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States